CLINICAL TRIAL: NCT06608927
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter, Phase 3 Trial of Quemliclustat and Chemotherapy Versus Placebo and Chemotherapy in Patients With Treatment-Naive Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of Quemliclustat and Chemotherapy Versus Placebo and Chemotherapy in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: PRISM-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRISM-1; 2024-513317-12-00 (EU CTIS Number); jRCT2061240084 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Quemliclustat; CD73 Inhibitor; Metastatic Pancreatic Ductal Adenocarcinoma; Treatment naive; Pancreatic cancer; PRISM-1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — quemliclustat; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental Arm) (Experimental): Quemliclustat, nab-paclitaxel and gemcitabine will be administered by IV infusion
  Interventions: Drug: Quemliclustat; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm B (Comparator Arm) (Placebo Comparator): Placebo, nab-paclitaxel and gemcitabine will be administered by IV infusion
  Interventions: Drug: Placebo; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Quemliclustat — Administered as specified in the treatment arm
  Arms: Arm A (Experimental Arm)
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Arm B (Comparator Arm)
Drug: Nab-paclitaxel — Administered as specified in the treatment arm
Drug: Gemcitabine — Administered as specified in the treatment arm

SUMMARY:
The purpose of this study is to compare overall survival of quemliclustat, nab-paclitaxel and gemcitabine versus placebo, nab-paclitaxel and gemcitabine in all randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed PDAC that is metastatic.
* Have not been previously treated for PDAC in the metastatic setting.

  1. Prior neoadjuvant and/or adjuvant therapy for PDAC is permitted if completed at least 12 months before randomization.
  2. Prior palliative radiotherapy is allowed if completed at least 2 weeks prior to randomization and AEs have resolved to Grade 1 or less before randomization.
  3. Prior and/or placement of a biliary stent/tube is permitted if any treatment-related AEs have improved to Grade ≤ 1 and the patient is not exhibiting any signs/symptoms of biliary obstruction.
* Eastern Cooperative Oncology Group PS of 0 to 1.
* At least 1 target lesion measurable by computed tomography (CT)/magnetic resonance imaging (MRI) per RECIST v1.1. not within a field of prior radiation therapy.

Exclusion Criteria:

* Previously treated for locally advanced, unresectable PDAC.
* History of brain metastases or leptomeningeal metastases.
* Prior treatment with a CD73 antagonist or inhibitor.
* Underlying medical conditions that, in the investigator or sponsor's opinion, will make the administration of study-specified therapy hazardous

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 72 months

SECONDARY OUTCOMES:
Progression-free Survival (PFS) as determined by the Investigator according to RECIST v1.1 | Up to 72 months
Objective response rate (ORR) as determined by the Investigator according to RECIST v1.1 | Up to 72 months
Duration of response (DoR) as determined by the Investigator according to RECIST v1.1 | Up to 72 months
Disease Control Rate (DCR) as determined by the Investigator according to RECIST v1.1 | Up to 72 months
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (125):
- United States (49):
  - Mayo Clinic Arizona - Phoenix Campus, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Diego Health, La Jolla, California
  - Cancer & Blood Specialty Clinic - Los Alamitos, Los Alamitos, California
  - Keck Medicine of USC - Keck Hospital of USC, Los Angeles, California
  - Sutter Medical Center, Roseville, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA Health - Santa Monica Cancer Care, Santa Monica, California
  - USOR - Rocky Mountain Cancer Centers - Denver - Midtown, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - USOR - Illinois Cancer Specialists - Arlington Heights, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Cancer Center of Kansas - Medical Arts Tower, Wichita, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Cancer & Hematology Centers of Western Michigan - Lemmen-Holton Cancer Pavilion, Grand Rapids, Michigan
  - HealthPartners Cancer Research Center - Cancer Center at Regions Hospital, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - MediSync Clinical Research - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York University Medical Oncology Associates, New York, New York
  - Columbia University Irving Medical Center - Herbert Irving Pavilion, New York, New York
  - Memorial Sloan-Kettering Cancer Center - New York - Rockefeller Outpatient Pavilion, New York, New York
  - Mount Sinai Medical Center Comprehensive Cancer Center, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - USOR - Texas Oncology - Austin Midtown, Austin, Texas
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - USOR - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - USOR - Texas Oncology - Deke Slayton Cancer Center, Webster, Texas
  - Inova Medical Group - Hematology Oncology - Arlington, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Summit Cancer Centers - Spokane Valley, Spokane, Washington
  - USOR - Northwest Cancer Specialists, P.C. dba Compass Oncology - Vancouver Cancer Center, Vancouver, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - Monash Health, Clayton
  - Oncology West - Murdoch, Murdoch
  - Wollongong Hospital, Wollongong
- Austria (4):
  - Salzburg Cancer Research Institute, Salzburg
  - Universitätsklinikum Sankt Pölten, Sankt Pölten
  - Krankenhaus Der Barmherzigen Brüder Wien, Vienna
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - Imeldaziekenhuis, Bonheiden
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk
- Canada (4):
  - Ottawa Hospital - General Campus, Ottawa
  - Hôtel-Dieu de Sherbrooke, Sherbrooke
  - Princess Margaret Cancer Centre, Toronto
  - Sunnybrook Health Sciences Centre - Bayview Campus, Toronto
- Czechia (3):
  - Fakultni Nemocnice Brno, Brno
  - Nemocnice AGEL Nový Jičín a.s., Nový Jičín
  - Fakultni nemocnice v Motole, Prague
- France (5):
  - Centre Georges François Leclerc, Dijon
  - Hôpital Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Gustave Roussy, Villejuif
- Germany (10):
  - Katholisches Klinikum Bochum - St. Josef-Hospital, Bochum
  - Krankenhaus Nordwest, Frankfurt am Main
  - Facharztzentrum Eppendorf, Hamburg
  - Katholisches Marienkrankenhaus, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn - Klinikum am Gesundbrunnen, Heilbronn
  - Otto-von-Guericke Universität, Magdeburg
  - Elblandklinikum Riesa, Riesa
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Italy (12):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Ospedale di Cremona, Cremona
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero - Universitaria di Modena, Modena
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Ospedale Guglielmo da Saliceto, Piacenza
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero Universitaria Delle Marche, Torrette
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (7):
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of JFCR, Kōtō City
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
  - National Cancer Center Hospital, Tokyo
  - Toyama University Hospital, Toyama
  - Yamaguchi University Hospital, Ube
  - Kanagawa Cancer Center, Yokohama
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Cha Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (12):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Institut Català d'Oncologia Girona (ICO Girona), Girona
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Alvaro Cunqueiro - Clinico Universitario Vigo, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Hull University Teaching Hospitals NHS Trust, Cottingham
  - Royal Free London NHS Foundation Trust, London
  - Sarah Cannon Research Institute London, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy/

REFERENCES:
- See also: PRISM-1 - Public website — https://trials.arcusbio.com/study/?id=PRISM1